CLINICAL TRIAL: NCT04180826
Title: Impact of Verticalization on Intracranial Hemodynamics Assessed by Continuous Transcranial Doppler Monitoring at the Acute Phase of Ischemic Stroke
Brief Title: STAND: iSchemic sTroke evAluated at Bed Side With ultrasouND
Acronym: STAND
Status: Terminated | Type: Observational
Why Stopped: alll patients have been included
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Collaborators: Hopital Lariboisière (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A03454-51
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Ischemic Stroke; Carotid Stenosis
MeSH Terms: conditions — Ischemic Stroke; Carotid Stenosis | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stenosis: Patients with stenosis
  Interventions: Other: Observational
- No stenosis: Patients without stenosis
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Initially, the patient will be placed in a strict supine position (at 0°) in his hospital bed, according to the usual care.
  In a second step, the patient will be verticalized (from 0° to 90°). Intracranial hemodynamics parameters in supine position and during verticalization will be continuously recorded by attaching the ATYS TCD-X® transcranial Doppler helmet attached with glasses.
  After 15 minutes of recording, the patient will be placed back in supine position. The end of the patient's participation in the study will correspond to the removal of the ATYS TCD-X® helmet.

SUMMARY:
Ischemic strokes account for more than 80% of strokes. Ischemic strokes are caused by the occlusion of an intracranial artery by a thrombus, responsible for tissue ischemia related to a decrease in local cerebral blood flow (CBS). Thus, the management of patients with Ischemic strokes is based on the preservation of an area that maintains sufficient intracranial hemodynamics (IH) and achieves the fastest possible recanalization. The impact of the patient's position (supine or seated position) on the IH in the event of narrowing or occlusion of an artery is poorly assessed but may be of particular importance. In practice, variations in blood flow according to the positioning of the patient's body can be measured using a transcranial Doppler. It is a simple, non-invasive and painless examination that provides the patient's bed with data on the intracerebral hemodynamic profile of patients.

This study was implemented because there are no studies known to us that evaluate the effect of verticalization on intracerebral hemodynamics based on the presence of upstream arterial stenosis or occlusion and other multimodal evaluation data in transcranial Doppler.

ELIGIBILITY:
Inclusion criteria

* Patient over 18 years of age
* acute ischemic stroke or transient ischemic attack
* symptoms onset < 48 hours
* Absence of homolateral or downstream intracranial stenosis or M1 occlusion
* Verticalization authorized by the referent clinician.
* Rankin's score before AIC/AIT ≤ 2
* Non-opposition to participation in the study

Criteria for inclusion of cases

- Carotid stenosis of more than 50% NASCET or an occlusion

Criteria for including witnesses - Absence of carotid stenosis greater than 50% NASCET or occlusion

Criteria for non-inclusion

- Disrupted vigilance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with ischemic stroke or transient ischemic attack of less than 48 hours with or without carotid stenosis greater than 50% NASCET or occlusion
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Change in the monitoring of patient care | 2 minutes after verticalization
  drop of more than 10% of the mean velocity between the supine and seated position

CONTACTS AND LOCATIONS:
Locations (1):
- Mikaël Mazighi, Paris, France

IPD SHARING:
Plan to Share IPD: No